CLINICAL TRIAL: NCT00540631
Title: A Multicentre Randomized Placebo-controlled Double-blind Clinical Trial for Evaluation of Safety and Efficacy of a Specific Immunotherapy With an Aluminium Hydroxide-adsorbed Allergoid Preparation of House Dust Mite (Dermatophagoides Pteronyssinus) in Patients With Rhinitis/Rhinoconjunctivitis and/or Allergic Asthma Bronchiale
Brief Title: Multicenter Trial of Immunotherapy With House Dust Mite Allergoid
Acronym: ACRI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL0106ac; 2006-000934-11 (EudraCT Number)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Rhinoconjunctivitis
Keywords: House Dust Mite Allergen; Aluminium hydroxide-adsorbed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P (No Intervention): subcutaneous treatment with placebo Placebo- physiological saline containing histamine-dihydrochloride 0.1mL, 0.2mL, 0.4mL, 0.6mL of strength A(1000TU/mL) followed by 0.1mL, 0.4mL, 0.6mL by strength B (10000TU/mL) in weekly intervals
- A (Experimental): Active treatment with house dust mite extract
  Interventions: Biological: specific immunotherapy with Acaroid, subcutaneously, Up-titration till strength B 0.6 mL (6000 TU)

INTERVENTIONS:
Biological: specific immunotherapy with Acaroid, subcutaneously, Up-titration till strength B 0.6 mL (6000 TU) — Injection Number Date Proposed Dose Individual Dose Strength A=1000 TU/ml B=10000TU/ml ml Dose per Injection
  1. to be det. A 0.1 100 TU
  2. 7 (+7) days later A 0.2 200 TU
  3. 7 (+7) days later A 0.4 400 TU
  4. 7 (+7) days later A 0.6 600 TU
  5. 7 (+7) days later B 0.1 1000 TU
  6. 7 (+7) days later B 0.2 2000 TU
  7. 7 (+7) days later B 0.4 4000 TU
  8. 7 (+7) days later B 0.6 6000 TU
  Maintenance (Init 2,4) 4-6 weekly B 0.6 6000 TU To be continued Injection Number Date Proposed Dose Individual Dose Strength A=1000 TU/ml B=10000TU/ml ml Dose per Injection
  1. to be det. A 0.1 100 TU
  2. 7 (+7) days later A 0.2 200 TU
  3. 7 (+7) days later A 0.4 400 TU
  4. 7 (+7) days later A 0.6 600 TU
  5. 7 (+7) days later B 0.1 1000 TU
  6. 7 (+7) days later B 0.2 2000 TU
  7. 7 (+7) days later B 0.4 4000 TU
  8. 7 (+7) days later B 0.6 6000 TU
  Maintenance (Init 2,4) 4-6 weekly B 0.6 6000 TU To be continued
  Arms: A

SUMMARY:
Multicenter Immunotherapy House Dust Mite Allergoid

DETAILED DESCRIPTION:
A multicentre randomized placebo-controlled double-blind clinical trial for evaluation of safety and efficacy of a specific immunotherapy with an aluminium hydroxide-adsorbed allergoid preparation of house dust mite (Dermatophagoides pteronyssinus) in patients with rhinitis/rhinoconjunctivitis and/or allergic asthma bronchiale

ELIGIBILITY:
Inclusion Criteria:

* Positive SPT
* Positive EAST
* Positive specific provocation test

Exclusion Criteria:

* Serious chronic diseases
* other perennial allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change of the area under the curve (AUC)of the Symptom-Medication-Score (SMS)after 2 years of double-blind treatment to baseline | November 2007 - February 2010

SECONDARY OUTCOMES:
Change of the AUC of the SMS after one year to baseline. | 1 year
Change of Nasal Eosinophil Cationic Protein (ECP) after 2 years to baseline | 2 years
Immunologic changes IgE, IgG1 and IgG4 | 2 years
Tolerability and safety of treatments during the entire study period | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Riechelmann, MD, Principal Investigator — University Ulm, Germany
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- See also: leader in specific allergy research and therapy — http://www.allergopharma.de